CLINICAL TRIAL: NCT02067143
Title: National Treatment Program of Philadelphia Chromosome-negative Adult Acute Lymphoblastic Leukemia With Pegylated Asparaginase Added to a Lineage-Targeted Risk- and Minimal Residual Disease-Oriented Strategy
Brief Title: MRD/Risk-oriented Therapy of Adult Ph- ALL Including Pegylated Asparaginase and Lineage-targeted Methotrexate
Acronym: LAL1913
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1913
Record Dates: First submitted 2014-02-17; First posted 2014-02-20 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Untreated Philadelphia Positive Acute Lymphoblastic Leukemia; De Novo; Secondary; Low-dose Corticosteroids Pretreatment
Keywords: Untreated philadelphia positive acute lymphoblastic leukemia; De novo; Secondary; Low-dose corticosteroids pretreatment; Pegylated asparaginase; Lineage-targeted risk and minimal residual disease
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasm, Residual | interventions — aspartyl-aspartic acid; Cytarabine; Mercaptopurine; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study population (Experimental): In this phase II multicentric trial, eligible patients with Ph- ALL/LL will receive homogeneous supportive care and chemotherapy and will be homogeneously analyzed for response at prefixed timepoints from induction day 1. For risk-/MRD-oriented therapy, CR patients will be stratified by risk class according to diagnostic characteristics, MRD study and CT/PET (LL only) results during early consolidation.
  Interventions: Drug: Prephase PDN + CY; Drug: Cycle 1 Induction; Drug: Cycle 2 Induction / Early consolidation; Drug: Cycle 3 Early consolidation; Drug: Cycle 4 Consolidation; Drug: Cycle 5 Consolidation; Drug: Cycle 6 Consolidation; Drug: Cycle 7 Consolidation; Drug: Cycle 8 Reinduction; Drug: Maintenance; Procedure: Allogeneic SCT or Autologous SCT

INTERVENTIONS:
Drug: Prephase PDN + CY
Drug: Cycle 1 Induction
  Other Names: VCR + IDR + DXM + ASP + IT
Drug: Cycle 2 Induction / Early consolidation
  Other Names: IDR + CY + ARA-C + ASP + 6MP + DXM + IT
Drug: Cycle 3 Early consolidation
  Other Names: MTX + ARA-C
Drug: Cycle 4 Consolidation
  Other Names: VCR + IDR + CY + ARA-C + 6-MP + DXM + IT
Drug: Cycle 5 Consolidation
  Other Names: MTX + ASP + 6-MP
Drug: Cycle 6 Consolidation
  Other Names: VCR + IDR + CY + ARA-C + ASP + 6MP + DXM + IT
Drug: Cycle 7 Consolidation
  Other Names: MTX + ARA-C
Drug: Cycle 8 Reinduction
  Other Names: VCR + IDR + DXM + PDN + CY + IT
Drug: Maintenance — If MRD negative MRD u/k SR
  Other Names: CY or VP and 6MP/MTX + 12 cycles of 6MP/MTX
Procedure: Allogeneic SCT or Autologous SCT — If MRD positive MRD u/k HR
  Other Names: + Maintenance

SUMMARY:
This study will be conducted in different centres and will study adult patients with Philadelphia chromosome-negative (Ph-) acute lymphoblastic leukemia (ALL). The study treatment will include a induction/consolidation therapy incorporating pegylated Asparaginase (Peg-ASP) and lineage-targeted high-dose methotrexate plus other antileukemic drugs, for the achievement of an early negative minimal residual disease (MRD) status. The MRD study supports a risk/MRD-oriented final consolidation phase.

DETAILED DESCRIPTION:
The aim of this clinical study in adult ALL is to improve , by risk category, the overall disease-free survival in relation to the achievement of an early MRD negative status and following induction/consolidation with Peg-ASP, lineage-targeted methotrexate infusions and other disease-specific therapeutic elements, with or without the application of allogeneic or autologous SCT depending on risk class and MRD study results. A survey of severe infections occurring along the entire chemotherapy and stem cell transplant program and until 2 years from the achievement of CR will be performed with the aim to increase the knowledge of these complications and to evaluate their impact on the antileukemic program and on the long term outcome of the underlying malignancy. The prospective survey of severe infections will be performed as an ancillary observational objective of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws.
* Age 18-65 years.
* A diagnosis of untreated Ph- ALL or LL is required, either de novo or secondary to chemo-radiotherapy for other cancer. Pretreatment with low-dose corticosteroids in patients presenting with hyperleukocytosis is allowed. All diagnostic procedures need to be performed on freshly obtained bone marrow (BM) and peripheral blood (PB) samples. The diagnosis must be one of: de novo ALL, secondary ALL, B-/T-cell LL Full cytological, cytochemical, cytogenetic and immunobiological disease characterization according to EGIL and WHO classifications. Bone marrow and peripheral blood sampling (ALL) or biopsy specimen (LL) are required for MRD study. Detailed indications on patient registration, storage of representative diagnostic material and diagnostic work-up, including the forwarding of samples for MRD study are given in Appendix B.
* Bone marrow and peripheral blood sampling (ALL) or biopsy specimen (LL) for MRD study.
* ECOG performance status 0-2, unless a performance of 3 is unequivocally caused by the disease itself and not by preexisting comorbidity, and is considered and/or documented to be reversible following the application of antileukemic therapy and appropriate supportive measures.

Exclusion Criteria:

* Diagnosis of Burkitt's leukemia or lymphoma.
* Down's syndrome
* Pre-existing, uncontrolled pathology such as heart failure (congestive/ischemic, acute myocardial infarction within the past 3 months, untreatable arrhythmias, NYHA classes III and IV), severe liver disease with serum bilirubin >3 mg/dL and/or ALT >3 x upper normal limit (unless attributable to ALL), kidney function impairment with serum creatinine >2 mg/dL (unless attributable to ALL), and severe neuropsychiatric disorder that impairs the patient's ability to understand and sign the informed consent, or to cope with the intended treatment plan. N.B. For altered liver and kidney function tests, eligibility criteria can be reassessed at 24-96 hours, following the institution of adequate supportive measures.
* Pre-existing HIV positive serology (i.e. already known before enrolment). If HIV positivity is detected after enrolment, the patient is sent off study.
* A history of cancer that is not in a remission phase following surgery and/or radiotherapy and/or chemotherapy, with life expectancy <1 year.
* Pregnancy declared by the patient herself, unless a decision is taken with the patient to induce a therapeutic abortion in order to carry on with ALL therapy. A pregnancy test is performed at diagnosis but does not preclude the enrolment into study. Fertile patients will be advised to adopt contraceptive methods while on treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-05-20 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Number of patients on disease free survival (DFS). | At two years.
  DFS is defined as the time interval between the evaluation of CR and relapse of the disease or death in first Complete Response (CR); patients still alive, in first CR, will be censored at the time of the last follow-up. In this case, the DFS will be truncated at 2 years.

SECONDARY OUTCOMES:
The rate of patients in complete remission (CR). | After approximately two months from start of treatment.
The rate of early bone marrow MRD negativity. | At 4 timepoints (week 4, 10, 16 22).
Early bone marrow MRD response (<10-4). | At 4 weeks following induction cycle 1 with Peg-ASP.
Overall Survival (OS) estimation. | At two years from diagnosis.
Cumulative Incidence of Relapse (CIR) estimation. | At two years from CR achievement.
The rate of patients dead due Treatment-related mortality (TRM). | By the end of the study (4.5 years from first centre opened).
Composite DFS, OS, CIR. | At two years from CR achievement and rate of TRM in LL patients.
Description of Minimal Residual Disease (MRD) monitoring. | During treatment at time point 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12.
Number of Severe Infections (SI) during treatment. | At the end of the study (4.5 years from first centre opened).
  Description: Number and type.
Rate of Adverse Events (AE). | By the end of the study (4.5 years from first centre opened)
  Excluding SI.
Composite evaluation of impact of age (≤55 and >55) and risk category group (SR, HR, VHR - as defined) on outcomes: DFS, CIR. | At two years for CR achievement, OS at two years from diagnosis and TRM.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, Pr., Study Chair — Azienda ULSS 12 Veneziana; Roberto Foà, Pr., Study Director — Policlinico Umberto I, Hematology Department.
Locations (61):
- Italy (61):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - Az.Ospedaliera S.G.Moscati, Avellino
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Azienda Ospedaliera - Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Comprensorio Sanitario di Bolzano - Azienda Sanitaria dell'Alto Adige - Ematologia e Centro TMO - Ospedale S.Maurizio, Bolzano
  - Spedali Civili - Brescia - Azienda Ospedaliera - U.O. Ematologia, Brescia
  - Divisione di Ematologia Ospedale A. Perrino, Brindisi
  - Ao Brotzu, Presidio Ospedaliero A. Businco - Cagliari - Sc Ematologia E Ctmo, Cagliari
  - CTMO - Ematologia - Ospedale "Binaghi", Cagliari
  - Unità Operativa Complessa di Onco-Ematologia - A.O. S.Anna e S.Sebastiano, Caserta
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Cona
  - Sezione di Ematologia C.T.M.O. Istituti Ospitalieri, Cremona
  - S.C. Ematologia ASO S. Croce e Carle, Cuneo
  - IRCCS_AOU San Martino-IST.Clinica Ematologica, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte" P.O. Papardo, Messina
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - Azienda Ospedaliera "S.Gerardo", Monza
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - U.O. CTMO Ematologia - Osp. S.Francesco, Nuoro
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto Dipart. Biomedico di Medicina Interna - A.U. Policlinico "Paolo Giaccone", Palermo
  - Casa Di Cura La Maddalena S.P.A. - Dipartimento Oncologico Di Iii Livello - Palermo - Uo Oncoematologia E Tmo, Palmero
  - Day Hospital dell'U.O.C di Ematologia e CTMO Padiglione 1 TORRE DELLE MEDICINE, 6° piano, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Sezione di Ematologia ed Immunologia Clinica - Ospedale S.Maria della Misericordia, Perugia
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Ematologia - Ospedale San Carlo, Potenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Sezione di Ematologia Cancer Center Humanitas, Rozzano
  - UOC di Ematologia e Trapianti di Cellule Staminali Emopoietiche - AOU San Giovanni di Dio e Ruggi D'Aragona, Salerno
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Dipartimento di Oncologia ed Ematologia S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Ospedale Mauriziano Umberto I - Torino - Scdu Ematologia, Torino
  - U.L.S.S. 9 UOC Ematologia - Ospedale Ca' Foncello, Treviso
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari Azienda Ospedaliero-Universitaria, Udine, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bassan R, Chiaretti S, Della Starza I, Spinelli O, Santoro A, Paoloni F, Messina M, Elia L, De Propris MS, Scattolin AM, Audisio E, Marbello L, Borlenghi E, Zappasodi P, Mauro E, Martinelli G, Mattei D, Fracchiolla N, Bocchia M, De Fabritiis P, Bonifacio M, Candoni A, Cassibba V, Di Bartolomeo P, Latte G, Trappolini S, Guarini A, Vitale A, Fazi P, Piciocchi A, Rambaldi A, Foa R. Pegaspargase-modified risk-oriented program for adult acute lymphoblastic leukemia: results of the GIMEMA LAL1913 trial. Blood Adv. 2023 Aug 22;7(16):4448-4461. doi: 10.1182/bloodadvances.2022009596. PMID 37276451
- [Derived] Piciocchi A, Messina M, Elia L, Vitale A, Soddu S, Testi AM, Chiaretti S, Mancini M, Albano F, Spadano A, Krampera M, Bonifacio M, Cairoli R, Vetro C, Colella F, Ferrara F, Cimino G, Bassan R, Fazi P, Vignetti M. Prognostic impact of KMT2A-AFF1-positivity in 926 BCR-ABL1-negative B-lineage acute lymphoblastic leukemia patients treated in GIMEMA clinical trials since 1996. Am J Hematol. 2021 Sep 1;96(9):E334-E338. doi: 10.1002/ajh.26253. Epub 2021 Jun 9. No abstract available. PMID 34048072
- See also: GIMEMA Foundation — http://www.gimema.it